CLINICAL TRIAL: NCT04871139
Title: Contrast-Enhanced Mammography (CEM) for the Evaluation and Targeted Biopsy of Suspicious Mammographic Architectural Distortions
Brief Title: An Imaging Technology, Contrast-Enhanced Mammography, in Predicting Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0031; NCI-2021-03404 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0031 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (iodine-based contrast, CEM) (Experimental): Patients receive iodine-based contrast agent IV and the undergo CEM over 10-15 minutes.
  Interventions: Procedure: Biopsy; Procedure: Contrast-Enhanced Mammography; Other: Questionnaire Administration; Other: Radioactive Iodine

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Contrast-Enhanced Mammography — Undergo CEM
  Other Names: CEM
Other: Questionnaire Administration — Ancillary studies
Other: Radioactive Iodine — Given IV

SUMMARY:
This clinical trial examines a new imaging technology, contrast-enhanced mammography, in predicting breast cancer. Contrast-enhanced mammography is similar to standard mammography, but it includes an intravenous (by vein) injection of iodine-based contrast, which makes tissue and blood vessels more visible in scans. Contrast-enhanced mammography may work better in detecting cancer in the breast that is not seen on other imaging tests and may help doctors find the most suspicious areas of the breast to biopsy, which could increase the chances of finding breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the added value of contrast enhancement of contrast-enhanced mammography (CEM) compared to full field digital mammography (FFDM) in predicting invasive malignancy or ductal carcinoma in situ (DCIS) in patients with suspicious mammographic architectural distortion (MAD)s.

SECONDARY OBJECTIVES:

I. To compare sensitivity, specificity, negative predictive value and positive predictive value of CEM versus FFDM, digital breast tomosynthesis (DBT), and ultrasound (US) in predicting invasive malignancy or DCIS in patients with suspicious MADs.

II. To evaluate whether the presence of enhancement on CEM correlates with the visibility of MAD on FFDM and DBT, or DBT only, and with the probability of malignancy.

III. To estimate the proportion of cases in which CEM changes the original target for a stereotactic biopsy.

IV. To evaluate the cancer detection rate and the outcomes (need for additional imaging, biopsies, and final pathologic results) of incidental CEM findings.

EXPLORATORY OBJECTIVES:

I. To evaluate the correlation of blood biomarkers and the presence of invasive cancer and DCIS on pathology in the study patients.

II. To evaluate the role of CEM enhancement pattern in choosing a precise target for a stereotactic biopsy.

III. To develop an objective method of quantifying the degree of enhancement above background using AI-based digital image analysis.

IV. To evaluate the technical feasibility of using CEM-guided or CEM-directed stereotactic biopsies in patients with suspicious MADs.

V. In patients who undergo CEM targeted or CEM directed biopsy we will evaluate the upgrade rate of DCIS to invasive malignancy or high-risk lesions to DCIS or invasive cancer for those patients who will require surgery as a part of their routine clinical care.

VI. To compare the performance of FFDM (obtained as a part of the recent prior screening or diagnostic mammographic work-up) and LE CEM images (obtained as a part of the CEM study) in terms of accuracy, sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) for the detection of invasive cancer and high-grade DCIS.

OUTLINE:

Patients receive iodine-based contrast agent intravenously (IV) and the undergo CEM over 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Women with suspicious MADs recommended for a stereotactic biopsy who underwent their diagnostic imaging work-up resulting in a biopsy recommendation at MD Anderson Cancer Center (MDACC) or at an outside facility with a technically acceptable quality of diagnostic mammography, and who are planning to have their biopsy at MDACC
* Age 25-85 years
* Willing to participate in the study, undergo an IV placement, able to undergo iodinated contrast injection, and able to provide informed consent

Exclusion Criteria:

* Reported history of an allergic reaction to iodinated contrast
* History of anaphylactic reaction to any substance
* Renal insufficiency
* Pregnancy or lactation within 6 months
* Breast surgery affecting the site of interest within prior 6 months
* Breast biopsy at the site of interest within the last 2 months

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of contrast-enhanced mammography (CEM) | Up to 3 years
  Will examine the accuracy of CEM compared to full field digital mammography (FFDM) in predicting invasive malignancy or ductal carcinoma in situ (DCIS) in patients with mammographic architectural distortion (MAD)s.

SECONDARY OUTCOMES:
Sensitivity of CEM, FFDM, digital breast tomosynthesis (DBT), and ultrasound (US) in predicting invasive malignancy or DCIS | Up to 3 years
  Will compare the sensitivity of CEM with that of FFDM, DBT, and US in predicting invasive malignancy or DCIS by using McNemar's test.
Specificity of CEM, FFDM, digital breast tomosynthesis (DBT), and US in predicting invasive malignancy or DCIS | Up to 3 years
  Will compare the specificity of CEM with that of FFDM, DBT, and US in predicting invasive malignancy or DCIS by using McNemar's test
Negative predictive value of CEM, FFDM, digital breast tomosynthesis (DBT), and US in predicting invasive malignancy or DCIS | Up to 3 years
Positive predictive value of CEM, FFDM, digital breast tomosynthesis (DBT), and US in predicting invasive malignancy or DCIS | Up to 3 years
Degree of enhancement on CEM | Up to 3 years
  Will examine the degree of enhancement on CEM and its correlation with the visibility of MAD on FFDM and DBT, or DBT only, and with the probability of malignancy.
Proportion of cases in which CEM changes the original target for a stereotactic biopsy | Up to 3 years
  We will estimate the proportion of cases in which CEM changes the original target along with an exact 95% confidence interval.
Cancer detection rate | Up to 3 years
  Will examine cancer detection rate and the outcomes (need for additional imaging, biopsies, and final pathologic results) of incidental CEM findings.

CONTACTS AND LOCATIONS:
Overall Officials: Olena Weaver, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org